CLINICAL TRIAL: NCT02529943
Title: Changes in Motor Latency During Spinal Decompression: Relationship to Outcomes
Status: Completed | Type: Observational
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Jonathan Norton, Ph.D., University of Saskatchewan
Other Study IDs: Norton15_05
Record Dates: First submitted 2015-08-13; First posted 2015-08-20 (Estimated); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Spinal Stenosis
Keywords: Spinal Stenosis; Motor Evoked Potential
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgery Group: Consecutive patients from a two surgeon practice

SUMMARY:
Is there a relationship between changes in motor evoked potential latency intraoperatively and post-operative changes in walking function in patients undergoing spinal decompression.

DETAILED DESCRIPTION:
Is there a relationship between changes in motor evoked potential latency intraoperatively and post-operative changes in walking function in patients undergoing spinal decompression. Tests will include the pre and post decompression MEP (motor evoked potential) latency and pre and post surgery walking speed and quality of life assessments.

ELIGIBILITY:
Inclusion Criteria:

* Central spinal stenosis
* Ability to ambulate prior to onset of symptoms

Exclusion Criteria:

* Arthritis affecting walking ability (hip, knee or ankle).
* Diabetes
* Implanted pacemaker or other electrostimulator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with central spinal stenosis scheduled for surgical decompression.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2016-05; Primary Completion 2021-10 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Motor Evoked Potential Latency | Day 0
  MEP latency at induction and completion of decompression

SECONDARY OUTCOMES:
10 m Timed Walking speed | pre-surgery and 3 months post surgery
  10m timed walk
Quality of Life measured in SF-36 | pre-surgery and 3 months post surgery
  SF-36

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Norton, PhD, Principal Investigator — University of Saskatchewan
Locations (1):
- Royal University Hospital, Saskatoon, Saskatchewan, Canada